CLINICAL TRIAL: NCT03661749
Title: Urinary Protein to Creatinine Ratio in Term Pregnant Women: What is the Effect of a Clean Catch Urine
Brief Title: Urinary Protein to Creatinine Ratio in Term Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Luke's Hospital, Pennsylvania (Other)
Responsible Party: Principal Investigator, James Anasti, MD, Clinical Professor of OB/GYN, St. Luke's Hospital, Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SLIR 2018-22
Record Dates: First submitted 2018-08-31; First posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Intervention Model Description: PR/CR urine collected by clean catch or non -clean catch technique will be compared in term pregnancy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clean catch (Experimental): women in this group will collect urine for PR/CR using a clean catch technique
  Interventions: Other: clean catch
- Non-clean catch (Placebo Comparator): women in this group will not employ clean catch technique
  Interventions: Other: clean catch

INTERVENTIONS:
Other: clean catch — clean catch technique applied to collect urine for PR/CR ratio

SUMMARY:
This study will determine the incidence of elevated U Pr/Cr in normal term pregnant women. In addition we will determine if a "clean catch" urine has an effect on the U Pr/Cr.

DETAILED DESCRIPTION:
Clean catch urine should be used due to possible vaginal secretion contamination with falsely elevated U Pr/Cr ratio. However, no supporting reference was found in the article and no control group with random urine collection for comparison to clean catch specimen U Pr/Cr was included in their study. The original studies that validated spot Pr/Cr urine as a predictor of 24 -hour total urine protein used random non-clean catch random urines . They had an r value of .93-.99 in estimating total protein excreted in 24 hours. At our institution we use Siemens-base test to determine U Pr/Cr. In the product insert the company states that no special patient preparation is necessary.

Thus, this study will determine the incidence of elevated U Pr/Cr in normal term pregnant women. In addition we will determine if a "clean catch" urine has an effect on the U Pr/Cr.

ELIGIBILITY:
Inclusion Criteria:

* women of 37 weeks gestation or greater

Exclusion Criteria:

* Urinary tract infections
* Hypertension
* Pre-eclampsia
* Renal dysfunction

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — pregnant females 37 weeks gestation or greater
Enrollment: 240 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
elevated PR/CR ratio using clean catch technique | through study completion, an average of 1 year
  this will be the proportion of patients with PR/CR ratio greater than or equal to 0.3 in urine using a clean catch method.

SECONDARY OUTCOMES:
Report the incident of PR/CR ratio greater than 0.3 | through study completion, average of 1 year
  overall incident of elevated PR/CR ratio in healthy term pregnant women

CONTACTS AND LOCATIONS:
Overall Officials: James N Anasti, MD, Principal Investigator — St Luke's University Hospital
Locations (1):
- St Luke's University Hospital, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided